CLINICAL TRIAL: NCT06808425
Title: Intervention With Weighted Blankets for Children With ADHD and Sleep Problems: Implementation and Effectiveness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Halmstad University (Other)
Responsible Party: Principal Investigator, Ingrid Larsson, RN, PhD, Professor, Professor, Halmstad University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F2024/38
Record Dates: First submitted 2025-01-29; First posted 2025-02-05 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-01

CONDITIONS: ADHD; Sleep Disturbances; Sleep; Sleep Problems
Keywords: implementation; sleep intervention; weighted blankets; children with ADHD; sleep problems
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Weighted blanket (Active Comparator)
  Interventions: Device: Intervention A
- Standard treatment (melatonin) (Active Comparator)
  Interventions: Drug: Intervention B

INTERVENTIONS:
Device: Intervention A — Weighted blanket
  Arms: Weighted blanket
Drug: Intervention B — Standard treatment (melatonin)
  Arms: Standard treatment (melatonin)

SUMMARY:
The aim is to study a sleep intervention with weighted blankets in children with ADHD and sleep problems regarding 1) short- and long-term effects on sleep and health-related outcomes in comparison with standard treatment (melatonin), 2) barriers and facilitators to implementation in routine clinical practice, and 3) health-economic outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with ADHD (DSM-5) and sleep problems (defined by screening instrument).
* Being a patient at child and adolescent mental health service (CAMHS) in Region Halland, Sweden.

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2034-02 (Estimated); Study Completion 2034-02 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Baseline, 1 month (m), 3 m, 6 m, 1 year, yearly for additional 9 years
  Insomnia Severity Index (ISI) assesses insomnia in the past two weeks by seven questions encompassing difficulties with 1) Sleep onset, 2) Sleep maintenance, and 3) Early morning awakening, as well as 4) Satisfaction with current sleep pattern, 5) Interference with daily functioning, 6) Noticeability of impairment attributed to the sleep problem, and 7) Level of distress caused by the sleep problem. Each question is assessed by a Likert scale. The answers is summed into a total score where a higher score indicates greater problems with insomnia.
Pediatric Insomnia Severity Index (PISI) | Baseline, 1 month (m), 3 m, 6 m, 1 year, yearly for additional 9 years
  Pediatric Insomnia Severity Index (PISI) is a parent-reported questionnaire assessing insomnia during the past week in children by six questions encompassing difficulties with 1) Sleep onset delay, 2) Sleep onset, 3) Nightly awakenings, 4) Falling back to sleep after nightly awakenings, 5) Daytime sleepiness, and 6) Sleep duration. The parents rate the frequency of sleep problems on scales, and the severity of sleep problems is summed into a total score, where a higher score indicates a greater degree of sleep problems.
Children's Sleep Habits Questionnaire (CSHQ) | Baseline, 1 month (m), 3 m, 6 m, 1 year, yearly for additional 9 years
  Children's Sleep Habits Questionnaire (CSHQ) - Swedish version (CSHQ-SWE) is a parent-reported questionnaire assessing sleep during the past week in children by 33 questions. The frequency of sleep problems or sleepiness during various activities for each question is estimated. The questions are divided into eight dimensions: 1) Bedtime resistance, 2) Sleep onset delay 3) Sleep duration, 4) Sleep anxiety, 5) Night wakings, 6) Parasomnias, 7) Sleep disordered breathing, and 8) Daytime sleepiness. The severity of sleep problems is summed into a total score, where a higher score indicates a greater degree of sleep problems.
Sleep Self Report (SSR) | Baseline, 1 month (m), 3 m, 6 m, 1 year, yearly for additional 9 years
  Sleep Self Report (SSR)2 is a questionnaire that assesses sleep-related difficulties with a focus on bedtime, sleep behavior and daytime sleepiness. The SSR contains 26 questions, of which 23 of the questions are answered by estimating frequency of events, and the remaining three questions are non-scored inquiries. The total score is summed up, with a higher score indicating more sleep problems.

SECONDARY OUTCOMES:
Child Outcome Rating Scale (CORS) | Baseline, 1 month (m), 3 m, 6 m, 1 year, yearly for additional 9 years
  Child Outcome Rating Scale (CORS) assesses everyday function and well-being in the domains of individual, family, school, and overall. Each domain is rated by the child on visual analogue scales, scored worst-best. A total score will also be utilized.
Outcome Rating Scale (ORS) | Baseline, 1 month (m), 3 m, 6 m, 1 year, yearly for additional 9 years
  assesses everyday function and well-being in the domains of individual, interpersonal, social role, and overall. Each domain is rated by the adult on visual analogue scales, scored worst-best. A total score will also be utilized.
Work and Social Adjustment Scale, Youth version (WSAS-Y) | Baseline, 1 month (m), 3 m, 6 m, 1 year, yearly for additional 9 years
  Work and Social Adjustment Scale, Youth version (WSAS-Y) assesses children's daily functioning. The instrument consists of five questions where children estimate the extent to which their problems affect school, daily skills, social activities, hobbies, and family and relationships. A total score is obtained, with higher scores indicating greater impact.
Work and Social Adjustment Scale, Parent version (WSAS-P) | Baseline, 1 month (m), 3 m, 6 m, 1 year, yearly for additional 9 years
  Work and Social Adjustment Scale, Parent version (WSAS-P) assesses children's daily functioning. The instrument consists of five questions where parents estimate the extent to which the children's problems affects school, daily skills, social activities, hobbies, and family and relationships. A total score is obtained, with higher scores indicating greater impact.
The Brief Child and Family Phone Interview (BCFPI) | Baseline, 1 month (m), 3 m, 6 m, 1 year, yearly for additional 9 years
  The Brief Child and Family Phone Interview (BCFPI) is a screening tool used to assess everyday functioning in children with neurodevelopmental conditions, as well as everyday functioning in the family. Selected scales from BCFPI will be utilized: "Impact on child functioning" (social participation, quality of social relations, and school participation and achievement), "Impact on family functioning" (family activities and family comfort), and "Parental functioning" (appetite problems, concentration problems, and emotional problems).
Lifestyle habits | Baseline, 1 month (m), 3 m, 6 m, 1 year, yearly for additional 9 years
  The child's height and weight, dietary habits (fruit intake, vegetable intake, consumption of sweets, and consumption of sugar-sweetened beverages), physical activity (fulfilling of recommendations, frequency of exercise during leisure time, and time spent on exercise during leisure time) and screen time and sedentary time (time spent in front of screen-based entertainment, time spent in sedentary gaming, and time spent using electronic devices for other purposes) are estimated by parents by selected questions included in the Health Behaviour in School-aged Children (HBSC) survey carried out by the Public Health Agency of Sweden.
The State-Trait Anxiety Inventory Scale - short form (Short STAI) | Baseline, 1 month (m), 3 m, 6 m, 1 year, yearly for additional 9 years
  The State-Trait Anxiety Inventory Scale - short form (Short STAI) assesses anxiety in children by six questions encompassing the themes of Calm, Tense, Upset, Relaxed, Content, and Worried. Each question is rated by the child, and the total score (best-worst) is obtained.
The Swanson, Nolan, and Pelham Scale - parent-reported version (SNAP-IV parent) | Baseline, 1 month (m), 3 m, 6 m, 1 year, yearly for additional 9 years
  The Swanson, Nolan, and Pelham Scale - parent-reported version (SNAP-IV parent) assesses ADHD symptoms and Oppositional Defiant Disorder (ODD) symptoms. The questionnaire includes 30 questions rated by the parent on a Likert scale. Attention deficit is covered by nine items, hyperactivity and impulsivity are combined and covered by nine items, and ODD is covered by eight items.The average rating per item may be calculated for the scales of attention deficit, hyperactivity and impulsivity, attention deficit/hyperactivity/impulsivity combined, and ODD. The additional four items are supplementary to ADHD (two items) and ODD (two items) and are not included in scoring. A higher score reflects greater severity of symptoms.
EQ-5D-Y-3L | Baseline, 1 month (m), 3 m, 6 m, 1 year, yearly for additional 9 years
  EQ-5D-Y-3L assesses health-related quality of life in children and adolescents. The questionnaire covers five domains: mobility, looking after myself, doing usual activities, having pain or discomfort, and feeling worried, sad or unhappy. Each domain is rated by the child on a Likert scale and answers are calculated into an index (worst-best). The questionnaire also includes a visual analogue scale (worst-best), reflecting current health state.
EQ-5D-3L | Baseline, 1 month (m), 3 m, 6 m, 1 year, yearly for additional 9 years
  EQ-5D-3L assesses health-related quality of life in adults. The questionnaire covers five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each domain is rated by the parent on a Likert scale and answers are calculated into an index (worst-best). The questionnaire also includes a visual analogue scale (worst-best), reflecting current health state.
Pain intensity | Baseline, 1 month (m), 3 m, 6 m, 1 year, yearly for additional 9 years
  Pain intensity during the last week is assessed by a visual analogue scale. The child estimates their perceived pain intensity during the last week on a scale between 0-100, where 0 corresponds to "no pain" and 100 corresponds to "worst imaginable pain".
Treatment Inventory Cost in Psychiatric Patients (TIC-P) | Baseline, 1 month (m), 3 m, 6 m, 1 year, yearly for additional 9 years
  Selected items from the Treatment Inventory Cost in Psychiatric Patients (TIC-P) will be utilized. TIC-P is a questionnaire that assesses absence from work and changes in work productivity for parents.
School absence and healthcare visits | Baseline, 1 month (m), 3 m, 6 m, 1 year, yearly for additional 9 years
  Parents will be asked to specify number of days their child has been absent from school and number of healthcare visits (specified by healthcare provider and healthcare professional) their child has made during the preceding month.

OTHER OUTCOMES:
Usage of weighted blanket and/or melatonin | Baseline, 1 month (m), 3 m, 6 m, 1 year, yearly for additional 9 years
  Parents will report frequency of usage of weighted blanket and/or melatonin on a 4-point scale (every night = 6-7 nights a week; almost every night = 4-5 nights a week; sometimes = 2-3 nights a week; almost never = 0-1 night a week). An additional three open-ended questions concerning how weighted blankets and/or melatonin have been used, the reason for usage, and thoughts about usage will be utilized.
Interviews with children and parents | 6 months and 1 year
  Individual interviews will be carried out with children and parents concerning the implementation of the intervention and the effect of the intervention, as well as how sleep affects child's everyday functioning, everyday activities, worry and anxiety, ADHD-related symptom burden, health-related quality of life, and sensory impressions.
Interviews with clinical staff | 6 months and 1 year
  Individual interviews and/or focus group interviews will be carried out with clinical staff concerning the implementation of the intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Halmstad University, Halmstad, Halland County, Sweden

IPD SHARING:
Plan to Share IPD: No